CLINICAL TRIAL: NCT00675493
Title: A Prospective, Multicentre, Open Label, Non-controlled, Observational, 24-week Study in Patients Using NovoMix® 30 (Biphasic Insulin Aspart 30) for Treatment of Type 1 and Type 2 Diabetes Mellitus in Romania
Brief Title: Observational Study of Type 1 and Type 2 Diabetes Patients Having Switched From Human Premixes to NovoMix®30
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-3567
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Start dose and frequency prescribed by the physician as a result of a normal clinical evaluation
  Other Names: NovoMix® 30

SUMMARY:
This trial is conducted in Europe. The aim of this observational study is to evaluate the blood glucose control (HbA1c) using NovoMix® 30 for treatment of type 1 and type 2 diabetes under normal clinical practice conditions in Romania.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 and type 2 diabetics who are treated with human premix insulin (the selection of the subjects will be at the discretion of the individual physician).

Exclusion Criteria:

* Subjects currently being treated with biphasic insulin aspart 30
* Subjects who were previously enrolled in this study
* Subjects with a hypersensitivity to biphasic insulin aspart 30 or to any of the excipients
* Women who are pregnant or have the intention of becoming pregnant within next 6 months
* Children below 10 years of age

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 1 and type 2 diabetes patients inadequately controlled on human premixes
Sampling Method: Non-Probability Sample
Enrollment: 942 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline | For the duration of the study

SECONDARY OUTCOMES:
Percentage of subjects achieving HbA1c below 7.0% and below or equal to 6.5% | after 12 weeks and 24 weeks of treatment
Change in FPG (glucose variability) | after 12 weeks and 24 weeks of treatment
Change in PPG (postprandial control) | after 12 weeks and 24 weeks of treatment
Change in insulin dose and number of injections | at 12 weeks and 24 weeks of treatment
Change in oral antidiabetic drug therapy | after 12 weeks and 24 weeks of treatment
Change in body weight | at 12 weeks and 24 weeks of treatment
Change in number of hypoglycaemic events | during 4 weeks proceeding routine visits at 12 weeks and 24 weeks of treatment
Number of adverse drug reactions (ADR) | after 12 weeks and 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Bucharest, Romania

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com